CLINICAL TRIAL: NCT00260559
Title: Outcomes After Esophagectomy With a Focus on Minimally Invasive Esophagectomy and Quality of Life
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, James Luketich, MD, University of Pittsburgh
Other Study IDs: STUDY20040382
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Esophagectomy; Esophageal Cancer
Keywords: Esophagectomy; Esophageal Cancer; Quality of Life; Minimally Invasive Esophagectomy; Laparoscopic Transhiatal Esophagectomy; Open Esophagectomy; Karnofsky Score; Dysphagia score; Heartburn Scale; Nutrition Score
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Questionnaires — Quality of life and heartburn assessment questionnaires are administered preoperatively and at set intervals postoperatively.

SUMMARY:
To assess short and long term outcomes after minimally invasive esophagectomy compared to open esophagectomy. To compare both standard outcome measures as well as patient derived outcome measures, in particular, quality of life (QOL). To look at the applicability of this QOL instrument to this patient group.

DETAILED DESCRIPTION:
Assess short and long term outcomes after minimally invasive esophagectomy(MIE) compared to open esophagectomy. Measure standard observer derived outcomes such as morbidity, mortality, tumor recurrence and also patient derived outcomes, in particular quality of life (QOL) using the MOS SF36 questionnaire. Evaluate whether the SF36 will accurately reflect pre and postoperative changes in clinical status in this patient group.Compare the results of this global QOL instrument (SF 36) to disease specific scales of dysphagia and reflux. Assess the impact of adjuvant or neoadjuvant therapy on QOL in this patient group and determine if any advantages of MIE can be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for MIE (Minimally Invasive Esophagectomy)
* Patients scheduled for open esophagectomy
* Signed informed consent

Exclusion Criteria:

* Patients who are unable to comprehend or complete the QOL instruments.
* Patients less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking surgical resection of their esophagus at the University of Pittsburgh Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 1999-05; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SF36 Quality of Life Questionnaire at 4 month postoperative | Baseline and 4 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 6 month postoperative | Baseline and 6 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 12 month postoperative | Baseline and 12 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 18 month | Baseline and 18 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 24 month | Baseline and 24 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 30 month | Baseline and 30 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.
Change from baseline in SF36 Quality of Life Questionnaire at 36 month | Baseline and 36 month postoperative
  The SF36 is an eight dimension Quality of Life Measurement. It provides two main Component scores, Physical Component Summary (PCS) and the Mental Component Summary (MCS). It includes 8 scales or sub-scores: Physical function (PF), role physical (RP), Bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MG). Each scale contributes a different amount to the component scores, which are calculated by a special algorithm that is licensed by Optum. The Component and sub-scales have a minimum of 0 and a maximum of 100. The higher the score represent the higher quality of life/less disability.

CONTACTS AND LOCATIONS:
Overall Officials: James D Luketich, MD, Principal Investigator — UPMC - Department of Cardiothoracic Surgery
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center - Department of Cardiothoracic Surgery, Pittsburgh, Pennsylvania
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No